CLINICAL TRIAL: NCT00432913
Title: The Effect of Two Dose Levels of Eicosapentaenoic Acid (EPA) on Apoptosis and Cell Proliferation in the Colonic Mucosa of Patients With a History of Colonic Polyps.
Brief Title: Effect of 2 Doses of EPA on Apoptosis and Cell Proliferation on Colon Mucosa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: S.L.A. Pharma AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPA/POL/02
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Adenomatous Polyps
Keywords: Eicosapentaenoic acid; EPA; EPA 99%; Fatty acid; omega-3; apoptosis; cell proliferation; colonic mucosa; polyps; adenomatous polyps; endoscopy; PUFA
MeSH Terms: conditions — Adenomatous Polyps; Hyperplasia; Polyps | interventions — Eicosapentaenoic Acid; Endoscopy; Colonoscopy; Clinical Chemistry Tests; Restraint, Physical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1g EPA per day (Active Comparator)
  Interventions: Drug: Eicosapentaenoic Acid (EPA); Procedure: Endoscopy; Procedure: Biopsies taken; Procedure: Clinical chemistry; Procedure: Haematology; Procedure: Physical examination; Procedure: Vital signs; Procedure: Urine pregnancy test; Procedure: Completion of patient diary card
- 2g EPA per day (Active Comparator)
  Interventions: Drug: Eicosapentaenoic Acid (EPA); Procedure: Endoscopy; Procedure: Biopsies taken; Procedure: Clinical chemistry; Procedure: Haematology; Procedure: Physical examination; Procedure: Vital signs; Procedure: Urine pregnancy test; Procedure: Completion of patient diary card
- Placebo (Placebo Comparator)
  Interventions: Procedure: Endoscopy; Procedure: Biopsies taken; Procedure: Clinical chemistry; Procedure: Haematology; Procedure: Physical examination; Procedure: Vital signs; Procedure: Urine pregnancy test; Procedure: Completion of patient diary card

INTERVENTIONS:
Drug: Eicosapentaenoic Acid (EPA) — Either 2 x 500mg EPA capsules in the morning and evening (2g per day EPA) or 1 x 500mg EPA and 1 x placebo in the morning and evening (1g per day EPA)
  Other Names: ALFA
  Arms: 1g EPA per day; 2g EPA per day
Procedure: Endoscopy — At baseline, month 3 and month 6.
  Other Names: Colonoscopy; Flexible sigmoidoscopy
Procedure: Biopsies taken — 9 biopsies taken for measurement of apoptosis (3 biopsies), cell proliferation (3 biopsies) and fatty acid levels (3 biopsies) at baseline, month 3 and month 6.
Procedure: Clinical chemistry — Full blood count at baseline, month 3 and month 6.
Procedure: Haematology — Urea and electrolytes, liver function tests, clotting profile and CRP at baseline, month 3 and month 6.
Procedure: Physical examination — Including cardio-respiratory and abdominal examination at baseline, month 3 and month 6.
Procedure: Vital signs — Height, weight, heart rate, blood pressure and temperature at baseline, month 3 and month 6.
Procedure: Urine pregnancy test — For subjects of child-bearing potential, urine pregnancy test at baseline, month 3 and month 6.
Procedure: Completion of patient diary card — Subjects are requested to complete when study medication is taken and in any new or unusual symptoms are experienced on a daily basis for 6 months.

SUMMARY:
The purpose of this study is to determine the effect of two doses purified EPA (an omega-3 fatty acid), on apoptosis (natural cell death) and cell proliferation (formation of new cells) in the lining of the colon for patients with a history of colonic polyps.

DETAILED DESCRIPTION:
Colorectal cancer is generally accepted to develop from changes within colonic adenomatous polyps. More than 90% of new large bowel cancers arise sporadically. The molecular events leading to the development of colorectal cancer from polyps are characterised by an imbalance in cell proliferation (formation of new cells) and apoptosis (natural cell death) from changes in the genes involved in normal colon cells.

Recent work at St George's Hospital Medical School, London, has shown significant beneficial effects on cell proliferation and apoptosis rates in the lining of the colon in subjects with a history of colonic adenomas using a highly purified, free-fatty acid form of eicosapentaenoic acid (EPA).

Comparator(s): 2g EPA per day for 6 months and 1g EPA per day for 6 months will be compared against placebo for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged over 18
* Patients of child-bearing potential must demonstrate a negative pregnancy test at screening, and should use a reliable form of contraception during the trial and for 1 month afterwards, e.g:
* Oral contraceptive + condom
* Intra-uterine device (IUD)+ condom
* Diaphragm with spermicide + condom
* Male partners of women of child bearing potential should use a reliable form of contraception during the trial and for 1 month afterwards, e.g:
* Oral contraceptive + condom
* Intra-uterine device (IUD)+ condom
* Diaphragm with spermicide + condom
* Patients must have a known history of colorectal adenomata and be under clinical follow-up for these, or be found to have one or more of these at the time of colonoscopy
* Patients must have provided written informed consent to participate

Exclusion Criteria:

* Patients who are allergic to fish
* Patients who have diabetes mellitus
* Patients who are pregnant or breast-feeding
* Patients taking aspirin or other non-steroidal anti-inflammatory drugs on a regular basis
* Patients who have aspirin-sensitive asthma
* Patients suffering from haemorrhagic disorders
* Patients who are taking warfarin or other anticoagulants
* Patients who have significant abnormalities on their screening blood tests
* Patients taking lipid lowering medication
* Patients with known inflammatory bowel disease (IBD), or previously unknown IBD until discovered at the time of their colonoscopy
* Patients with gastrointestinal malabsorptive disease
* Patients belonging to a known polyposis syndrome (e.g. FAP, HNPCC)
* Patients with a previous colonic resection for colorectal cancer
* Patients who are taking other fish-oil supplements (e.g. cod liver oil) who are unwilling to stop them for the duration of the study
* Patients who are deemed mentally incompetent, or have a history of anorexia nervosa or bulimia
* Patients with a history of alcohol or drug abuse, including laxative abuse
* Patients considered by their physician unlikely to be able to comply with the protocol.
* Patients who have taken part in an experimental drug study in the preceding 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To measure levels of apoptosis in the normal colonic mucosa in subjects with a history of colonic adenomas, before and after treatment with EPA 99%. | 3 months and 6 months
To measure levels of cell proliferation in the normal colonic mucosa in subjects with a history of colonic adenomas, before and after treatment with EPA 99%. | 3 months and 6 months

SECONDARY OUTCOMES:
To measure the tissue content of EPA in the colonic mucosa before, during and after treatment with EPA. | 3 months and 6 months
To determine the safety and tolerability of EPA. | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J West, MB BS FRCS, Principal Investigator — St. George's Hospital Medical School, London
Locations (2):
- S. Orsola Hospital, Bologna, Italy
- St. George's Hospital Medical School, London, United Kingdom